CLINICAL TRIAL: NCT03948100
Title: Dyadic Behavioral Interventions to Manage Physical Performance, Symptoms and Quality of Life for Patient Undergoing Radiotherapy and Their Family Caregivers
Brief Title: Dyadic Yoga Intervention in Improving Physical Performance and Quality of Life in Patients With Stage I-IV Non-small Cell Lung or Esophageal Cancer Undergoing Radiotherapy and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-0503; NCI-2018-03913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0503 (Other: M D Anderson Cancer Center); R37CA231522 (NIH)
Record Dates: First submitted 2019-04-05; First posted 2019-05-13 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Esophageal Carcinoma; Lung Non-Small Cell Carcinoma; Stage I Lung Cancer AJCC v8; Stage IA1 Lung Cancer AJCC v8; Stage IA2 Lung Cancer AJCC v8; Stage IA3 Lung Cancer AJCC v8; Stage IB Lung Cancer AJCC v8; Stage II Lung Cancer AJCC v8; Stage IIA Lung Cancer AJCC v8; Stage IIB Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8; Stage IVA Lung Cancer AJCC v8; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods; Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research staff blinded to group assignment will collect the assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (dyadic yoga) (Experimental): Patients and caregivers undergo dyadic yoga intervention session involving physical exercises and relaxation techniques over 60 minutes each for up to 15 sessions.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Yoga
- Group II (dyadic education) (Active Comparator): Patients and caregivers undergo dyadic education program session focusing on strategies of how to manage patient and caregiver symptoms over 60 minutes each for up to 15 sessions.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Undergo dyadic education program
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Group II (dyadic education)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Yoga — Undergo dyadic yoga
  Other Names: Yoga Therapy
  Arms: Group I (dyadic yoga)

SUMMARY:
This trial studies how well dyadic yoga intervention works in improving physical performance and quality of life in patients with stage I-IV non-small cell lung or esophageal cancer undergoing radiotherapy and their caregivers. Dyadic yoga intervention may help to improve physical function, fatigue, sleep difficulties, depressive symptoms, and overall quality of life for patients with non-small cell lung cancer and/or their caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To examine the extent to which the yoga program improves patient physical performance (i.e., 6-minute walk test [6MWT]) as compared to the education group.

SECONDARY OBJECTIVE:

I. To examine the extent to which the yoga program improves patient and caregiver quality of life (QOL) (SF-36) compared to the education group.

TERTIARY OBJECTIVES:

I. To explore if, compared to the education group, the yoga program improves symptom burden, reduces inflammatory cytokine and cortisol rhythmicity dysregulation, and improves dyadic symptom management skills at the end of treatment, which will in turn mediate intervention outcomes at the subsequent follow-up assessments.

II. To explore if baseline factors such as depressive symptoms moderate the treatment response. We also seek to explore if baseline factors such as depressive symptoms moderate the treatment response.

QUALITATIVE OBJECTIVE:

I. To understand the patient and caregiver experience of cancer, cancer treatment, and experience in the behavioral interventions, and explore emerging themes as possible mediators. We would also like to understand participants feedback on participating in this intervention via mobile application (app) delivery.

OUTLINE: Patients and caregivers are assigned to 1 of 2 groups.

GROUP I: Patients and caregivers undergo dyadic yoga intervention session involving physical exercises and relaxation techniques over 60 minutes each for up to 15 sessions.

GROUP II: Patients and caregivers undergo dyadic education program session focusing on strategies of how to manage patient and caregiver symptoms over 60 minutes each for up to 15 sessions.

After completion of study, patients and caregivers are followed up every 2 weeks for 3 months and then every month for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT ONLY: Diagnosed with stage I-IV non-small cell lung cancer (NSCLC) or esophageal cancer and going to receive at least 3 weeks of thoracic radiotherapy (RT)
* PATIENT ONLY: Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* PATIENT ONLY: Able to read, write and speak English
* PATIENT ONLY: Able to provide informed consent
* PATIENT ONLY: Having a family caregiver (e.g., spouse, sibling, adult child) who assists the patient during the cancer treatment (e.g., emotional support, transportation, meal preparation, care coordination, etc) per patient self-report. Note, patients must identify a family caregiver; however, the participation of the family caregiver is optional. For caregivers to be eligible, they must be at least 18 years old; able to read, write and speak English; and able to provide informed consent. Family caregivers may consent to participate in the intervention and caregiver assessments or only the assessments based on their preference.

Exclusion Criteria:

* PATIENT ONLY: Who have regularly (self-defined) participated in a mind-body practice in the year prior to diagnosis
* PATIENT ONLY: Patients who metastatic disease involving the central nervous system

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Patient 6-minute walk test (6MWT) | At 3 months post study
  Descriptive statistics for study variables and potential covariates will be computed and distribution characteristics of the variables will be examined. The difference between dyadic yoga (DY) and dyadic edication (DE) at 3 month follow-up (3MFU) will be tested at a two-sided .05 significance level.

SECONDARY OUTCOMES:
Patient and caregiver quality of life (QOL) | Up to 6 months post study
  Analyses will be similar to those for the primary outcome, except that we will use a dyadic model assuming additional dependence in outcomes between patient and caregiver outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Milbury, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Snyder S, Silva RF, Whisenant MS, Milbury K. Videoconferenced Yoga Interventions for Cancer Patients and their Caregivers during the COVID-19 Pandemic: A Report from a Clinician's Perspective. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211019111. doi: 10.1177/15347354211019111. PMID 34036820
- See also: MD Anderson Cancer Center — http://www.mdanderson.org